CLINICAL TRIAL: NCT04420910
Title: Investigation of Non-motor Symptoms, Balance, Muscle Strength, and Functional Mobility in Patients With Parkinson's Disease
Brief Title: Non-motor Symptoms, Balance, Muscle Strength, and Functional Mobility in Patients With Parkinson's Disease
Status: Completed | Type: Observational
Sponsor: Ankara Yildirim Beyazıt University (Other)
Responsible Party: Sponsor
Other Study IDs: 2019-71
Record Dates: First submitted 2020-06-04; First posted 2020-06-09 (Actual); Last update posted 2020-06-09 (Actual); Status verified 2020-06

CONDITIONS: Parkinson Disease; Balance; Muscle Strength; Mobility; Non-motor Symptoms
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Parkinson's disease group: being diagnosed with PD by a neurologist, being in Hoehn & Yahr Stage 1-3
  Interventions: Other: Non-Motor Symptoms; Other: Balance; Other: Lower Limb Strength; Other: Functional mobility
- Healthy group: 20 healthy volunteers with matching ages and genders.
  Interventions: Other: Non-Motor Symptoms; Other: Balance; Other: Lower Limb Strength; Other: Functional mobility

INTERVENTIONS:
Other: Non-Motor Symptoms — NMSs of the participants were evaluated using the Non-Motor Symptoms Scale (NMSS). The scale consists of 30 yes-no questions and is administered face to face with the therapist.
Other: Balance — To measure balance, the Biodex Balance System (Biodex Medical Systems, Shirley, NY, USA) was used. The participants were asked to position themselves in a comfortable position on the platform, and their foot position coordinates were recorded. The participants focused on a characteristic dot on the monitor screen. Their task was to balance the body in such a way that the dot was in the center of a circle displayed on the monitor at the point of intersection of the coordinate axes. The test consisted of three 20 s trials, each separated by 10 s breaks. Measurements were conducted while their eyes were open and close, and the results were analyzed by calculating the average value of the measurements.
Other: Lower Limb Strength — A Biodex® System 4 Dynamometer device was used to evaluate muscle strength. The participants' dominant extremity was determined by asking them the foot with which they most often hit the ball.The dynamometer arm of the device was placed at the lateral condyle level of the knee, and the belt at the distal end of the dynamometer was attached to the lower leg on the malleolus. Knee flexion and extension movements were evaluated in sitting position between 90ᵒ flexion and 0ᵒ extension angles. The individual was asked to perform it with the maximum strength, while the therapist motivated the individual with verbal stimulation.
Other: Functional mobility — The Timed Up and Go test (TUG) was used in the evaluation of functional mobility. . For this test, participants were seated on a standard armless chair and a cone was placed 3 meters away from the chair. Participants were instructed to stand up and (1) walk towards the cone, (2) turn around the cone, (3) walk back to the chair, and (4) sit back on the chair. It was stated that patients should walk without running but as fast as possible. Dual task performance was performed by adding cognitive and motor tasks into the TUG.

SUMMARY:
The purposes of this study is to examine balance, muscle strength, and mobility in relation with non-motor symptoms (NMSs) in patients with Parkinsosn's Disease (PD).

NMSs have been shown to be the key determinant of health-related quality of life (HRQoL) and have a greater effect on HRQoL compared to motor symptoms.Despite a growing literature on NMSs, there are few data on the association between NMSs and motor phenotypes of PD, and they have usually focused only on specific domains of NMSs, such as cognition, mood/anxiety issues, or sleep disorders.

When literature is examined, there is no study which examines balance, muscle strength, and mobility in relation with NMSs in patients with PD.For all these reasons, we think that balance, muscle strength, mobility, and NMSs in patients with PD are worse than those of the healthy individuals and that there is a relationship between NMSs and motor symptoms.

ELIGIBILITY:
Inclusion Criteria:

* being diagnosed with PD by a neurologist, being in Hoehn & Yahr Stage 1-3, having no musculoskeletal system problems in the previous 6 months, having a score of 24 or more in the Mini-Mental State Examination (MMSE), and being volunteer.

Exclusion Criteria:

* Healthy individuals of similar age and sex, without neurological problems, and who did not experience any musculoskeletal system problems in the previous 6 months were included in the control group.

Ages: 50 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: being diagnosed with PD by a neurologist, being in Hoehn & Yahr Stage 1-3 and healthy individuals of similar age and sex
Sampling Method: Probability Sample
Enrollment: 44 (Actual)
Dates: Start 2019-04-15 (Actual); Primary Completion 2019-08-15 (Actual); Study Completion 2019-09-15 (Actual)

PRIMARY OUTCOMES:
Non-Motor Symptoms | one hour
  Non-motor symptoms of the participants were evaluated using the Non-Motor Symptoms Scale (NMSS).Each item of the scale is scored between 0 and 30, with "yes" 1 point and "no" 0 point. According to the scoring result, "0" indicates no NMSs, "1-5" indicates mild NMSs, "6-9" indicates medium NMSs, "10-13" indicates heavy NMSs, and "≥14" indicates very heavy NMSs.
Balance | one hour
  To measure balance, the Biodex Balance System (Biodex Medical Systems, Shirley, NY, USA) was used.The test consisted of three 20 s trials, each separated by 10 s breaks. Measurements were conducted while their eyes were open and close, and the results were analyzed by calculating the average value of the measurements. As a result, overall stability and anteroposterior and mediolateral indexes were taken into account, and low values indicate high postural stability.
Lower limb strength | one hour
  A Biodex® System 4 Dynamometer device was used to evaluate muscle strength.Maximal concentric knee flexion and extension muscle strength was measured at 90 degrees/sec angular velocity with 5 repetition [19]. The flexion and extension peak torque (PT) values, peak torque/body weight (PT/BW) ratio, and hamstring/quadriceps (H/Q) ratio were recorded. Low values indicate decreased muscle strength.
Functional mobility | one hour
  The Timed Up and Go test (TUG) was used in the evaluation of functional mobility. Dual task performance was performed by adding cognitive and motor tasks into the TUG.. As the time increases, dual task performance decreases.

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara Yıldırım Beyazıt University, Faculty of Health Sciences,Department of Physiotherapy and Rehabilitation, Ankara, Esenboğa, Turkey (Türkiye)